CLINICAL TRIAL: NCT02579057
Title: Prospective, Randomized, Parallel-Group Pilot Study Comparing IV Furosemide to Subcutaneous Furosemide in Acute Decompensated Heart Failure Patients
Brief Title: Sub-Q Versus IV Furosemide in Acute Heart Failure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: scPharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00068019
Record Dates: First submitted 2015-10-14; First posted 2015-10-19 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Congestive Heart Failure
Keywords: Congestive heart failure; Furosemide
MeSH Terms: conditions — Heart Failure | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Furosemide Injection Solution, USP (Active Comparator): Single dose determined by Investigator (maximum dose 160mg) administered intravenously by IV bolus over approximately 2 minutes (reference treatment)
  Interventions: Drug: Furosemide Injection Solution, USP
- Furosemide Injection Solution (SCP-101) (Experimental): 80 mg dose administered subcutaneously as 30 mg over the first hour and then as 12.5 mg per hour over the subsequent 4 hours (test treatment)
  Interventions: Drug: Furosemide Injection Solution (SCP-101)

INTERVENTIONS:
Drug: Furosemide Injection Solution (SCP-101)
  Other Names: sc Furosemide
  Arms: Furosemide Injection Solution (SCP-101)
Drug: Furosemide Injection Solution, USP
  Other Names: IV furosemide
  Arms: Furosemide Injection Solution, USP

SUMMARY:
This study evaluates the clinical efficacy of subcutaneously administered Furosemide Injection Solution versus intravenous administration of Furosemide Injection, United States Pharmacopeia (USP) in adult patients presenting to a heart failure clinic with decompensated heart failure. Half of the patients will receive a subcutaneously administered Furosemide Injection Solution; the other half will receive an intravenous administration of Furosemide Injection.

DETAILED DESCRIPTION:
The prevalence of chronic heart failure is increasing, and despite advances in the treatment of chronic heart failure, in-hospital mortality and readmission are high. Heart failure costs the US about 32 billion per year, and a large percentage of the costs are due to hospitalizations. Most clinicians would agree that patients with decompensated heart failure presenting with hypotension, worsening renal function and altered mental status should be hospitalized. However, there is a subset of patients presenting with dyspnea and edema due to volume overload that necessitate rapid symptom improvement but are hemodynamically stable. Oral diuretics would likely be ineffective but hospital admission for IV diuretics seems excessive.

The research hypothesis is that subcutaneously administered furosemide will be an effective alternative to IV furosemide for hemodynamically stable chronic heart failure patients presenting with volume overload in the ambulatory setting. Patients will be randomized to receive Furosemide Injection, USP intravenously or Furosemide Injection Solution (SCP-101) delivered subcutaneously. The IV patients will get the usual care of the heart failure clinic, which includes having an IV placed and delivery of a one-time dose of IV furosemide with the dose determined by the providers (maximum dose 160mg IV). The subcutaneous patients will receive 80mg of Furosemide Injection Solution (SCP-101) administered subcutaneously over 5 hours (30mg in first hour and 12.5mg/hour for 4 hours).

Both groups of patients will be observed for 6 hours to assess diuresis. Patients will be asked to fill out a survey about their symptom improvement (Kansas City Cardiomyopathy questionnaire) and overall satisfaction related to the treatment experience. They will also be monitored for side effects including ototoxicity and discomfort at the access site (burning, itching, and pain). Electrolytes and renal function will be checked once after the patients receive diuretic therapy.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB) approved informed consent is signed and dated prior to any study-related activities.
* Male and female subjects > 18 years of age
* History of at least 3 months treated heart failure (NYHA class II/III/IV), or recent hospitalization for heart failure; presenting to Heart Failure Bridge Clinic (HFBC) with decompensated heart failure symptoms including elevated jugular venous pressure, dyspnea and peripheral edema where the decision is made to give IV diuretics
* Able to participate in the study in the opinion of the investigator
* Has the ability to understand the requirements of the study and is willing to comply with all study procedures

Exclusion Criteria:

* Presenting with symptoms where it is anticipated that there is a high chance of hospitalization such as ischemia, uncontrolled arrhythmia, infection, hemodynamic instability (elevated or low blood pressure), respiratory compromise, or electrolyte abnormalities (>25% increase in creatinine from baseline, potassium, hyponatremia).
* On experimental medication or currently participating in a cardiovascular research study.
* Presence or need for urinary catheterization, urinary tract abnormality or disorder interfering with urination
* Any surgical or medical condition which in the opinion of the investigator may interfere with participation in the study or which may affect the outcome of the study
* Inability to comply with study requirements

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Russell, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital Heart Failure Bridge Clinic, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Gilotra NA, Princewill O, Marino B, Okwuosa IS, Chasler J, Almansa J, Cummings A, Rhodes P, Chambers J, Cuomo K, Russell SD. Efficacy of Intravenous Furosemide Versus a Novel, pH-Neutral Furosemide Formulation Administered Subcutaneously in Outpatients With Worsening Heart Failure. JACC Heart Fail. 2018 Jan;6(1):65-70. doi: 10.1016/j.jchf.2017.10.001. Epub 2017 Dec 6. PMID 29226816

RESULTS

PARTICIPANT FLOW:
Groups:
- Furosemide IV: Single dose determined by Investigator (maximum dose 160mg) administered intravenously by IV bolus over approximately 2 minutes (reference treatment)
  Furosemide Injection Solution, United States Pharmacopeia (USP)
- Furosemide Subcutaneous (SC): 80 mg dose administered subcutaneously as 30 mg over the first hour and then as 12.5 mg per hour over the subsequent 4 hours (test treatment)
  Furosemide Injection Solution (SCP-101)
Period: Overall Study
Arm/Group | Furosemide IV | Furosemide Subcutaneous (SC)
Started | 19 | 21
Completed | 19 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Furosemide IV: Single dose determined by Investigator (maximum dose 160mg) administered intravenously by IV bolus over approximately 2 minutes (reference treatment)
  Furosemide Injection Solution, USP
- Total: Total of all reporting groups
Arm/Group | Furosemide IV | Furosemide Subcutaneous (SC) | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (13) | 59 (13) | 57 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 10 | 8 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 12 | 26
  White | 5 | 8 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 21 | 40
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 39.7 (11.2) | 37.8 (11.3) | 38.7 (11.2)
Ejection fraction [Median (Inter-Quartile Range); unit: % left ventricular function] | 20 [20 to 55] | 25 [15 to 55] | 25 [15 to 55]
Furosemide daily dose [Mean (Standard Deviation); unit: mg] | 228 (174) | 261 (164) | 246 (167)

OUTCOME MEASURES:

1. Primary Outcome: Urine Output
Description: The volume of urine produced in milliliters over the 6 hours after drug delivery will be measured.
Time Frame: 6-hour period
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Furosemide SC: 80 mg dose administered subcutaneously as 30 mg over the first hour and then as 12.5 mg per hour over the subsequent 4 hours (test treatment)
  Furosemide Injection Solution (SCP-101)
Arm/Group | Furosemide IV | Furosemide SC
Number analyzed (Participants) | 19 | 21
mL | 1636 (875) | 1515 (1000)

2. Secondary Outcome: Heart Failure Symptom Scoring/Symptom Improvement
Description: Will evaluate if subjective heart failure symptoms improve over the period of diuresis. Measured by Kansas City Cardiomyopathy Questionnaire
Time Frame: 6-hour period
Population: Data was not collected on enough patients to accurately analyze this endpoint. No data analysis was performed for this outcome.
Arm/Group | Furosemide IV | Furosemide SC
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Side Effects
Description: Cumulative total of pain, local skin reactions (including hematoma and induration) and electrolyte abnormalities.
Time Frame: Up to 6 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide IV | Furosemide SC
Number analyzed (Participants) | 19 | 21
Participants
  Hypokalemia | 0 | 1
  Skin irritation | 0 | 0
  Infusion site pain | 0 | 0

4. Secondary Outcome: Urine Sodium
Description: Total urinary sodium produced during the 6 hour urine collection
Time Frame: 6-hour period
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Furosemide IV | Furosemide SC
Number analyzed (Participants) | 19 | 21
mEq/L | 7.3 (35.3) | 32.8 (43.6)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Furosemide IV | Furosemide Subcutaneous (SC)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/19 | 1/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Furosemide IV (N=19) | Furosemide Subcutaneous (SC) (N=21)
Hypokalemia (General disorders) | 0 (0) | 1 (1) — Serum potassium < 3.5 mEq/L

LIMITATIONS AND CAVEATS:
This was a phase II exploratory trial with a small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT02579057/Prot_SAP_000.pdf